CLINICAL TRIAL: NCT01089842
Title: Randomized Clinical Trial to Assess the Efficacy and Cost-efficacy of Health Coaching to Promote Physical Activity in Secondary Prevention of Coronary Heart Disease
Brief Title: Health Coaching to Promote Physical Activity for Coronary Heart Disease Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Joan R Guma, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI08/90182; CIR08/034 (Other Grant/Funding Number: Institut Universitari Parc Taulí. Esfera UAB)
Record Dates: First submitted 2010-03-18; First posted 2010-03-19 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2010-02

CONDITIONS: Coronary Disease; Atherosclerosis
Keywords: Secondary Prevention; Health Promotion; Behavioral Medicine; Exercise Therapy
MeSH Terms: conditions — Coronary Disease; Atherosclerosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health coaching (Experimental)
  Interventions: Behavioral: Health coaching
- Control (No Intervention)
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Health coaching — Coaching based advice will be performed by previously trained nurses. Intervention will be directed to increase physical activity to achieve levels recommended on guidelines. Patients will receive one session per month during 6 months. Time for each session is estimated on 10 to 20 minutes. Sessions will be mostly carried out by phone, although physical attendance or internet services can also be used.
  Arms: Health coaching
Other: Usual care — Patients on control group will receive usual assistance, including physical activity counselling by their treating physician.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the efficacy of motivational interviewing-based coaching to increase physical activity to achieve guidelines recommendations for cardiovascular disease prevention.

DETAILED DESCRIPTION:
Cardiovascular diseases are the main cause of death in developed countries. Epidemiological studies have shown that a sedentary lifestyle is associated with an increased risk of cardiovascular diseases, mainly related to classical risk factors (obesity, diabetes, hypertension). International guidelines recommend, because of that, a minimum of 30 minutes per day at least 5 days per week of moderate physical activity for primary and secondary cardiovascular disease prevention.

Physical inactivity is an increasing public health problem in developed countries. It is known that clinical advice has a poor efficacy to increase levels of physical activity on individuals and new strategies need to be developed.

Coaching is a strategy of personal help that is being widely and successfully used in business world. It consists of an structured and individualized process of assistance to people to promote cognitive changes needed to achieve behavioural changes. It can be a complementary method to information and sanitary education emphasizing on consciousness and responsibility of the patient and is now starting to be used in medical practice. The purpose of the study is to define usefulness of an strategy based on coaching techniques to promote physical activity practice and healthy lifestyle on individuals with known coronary heart disease or cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients wiht coronary risk factors or known ischaemic heart disease defined as sedentary (<600MET-min/week).

Exclusion Criteria:

* Bundle branch block or pacemaker rhythm
* Limitation or contraindication to moderate physical activity (fast walking)
* Unstable clinical situation
* Communication difficulties due to language or sensorial deficiencies.
* Lack of informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-06 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Patients achieving recommended physical activity (>600 MET-minute/week) | 6 months
  Physical activity will be measured using the International Physical Activity Questionnaire (IPAQ)

SECONDARY OUTCOMES:
Cost-efficacy of coaching | 6 months
  Cost-efficacy will be measured using SF-12v2 quality of life questionnaire
Improvement on functional capacity | 6 months
  Exercise treadmill Bruce test will be used to assess cardiovascular fitness and compare functional capacity before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Joan R Guma, Principal Investigator — Corporacion Parc Tauli
Locations (1):
- Hospital de Sabadell, Sabadell, Barcelona, Spain